CLINICAL TRIAL: NCT00262574
Title: Phase 4 Study of Patients Receiving BNP or NTG (IV) During Angioplasty, Re-examined 24 Hours Later Using the Flow-mediated Brachial Artery Dilation Study, and Blood Assays for Pro BNP and ET1
Brief Title: Effect of BNP (Brain Natriuretic Peptides) on Endothelial Dysfunction Induced by Coronary Angioplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Baruch Padeh Medical Center, Poriya (Other Government)
Responsible Party: prof yonathan hasin, Israell health ministry
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20020474-Hasin-BNP.CTIL
Record Dates: First submitted 2005-12-06; First posted 2005-12-07 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2010-12

CONDITIONS: Coronary Artery Disease
Keywords: endothelial disfunction; BNP; PCI; coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Natriuretic Peptide, Brain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Nesiritide, — PCI

SUMMARY:
Patients receiving BNP or nitroglycerin (IV) during the angioplasty procedure. 24 h after the procedure, vascular reactivity will be re-examined using the brachial artery flow-mediated dilatation study. Blood assays for ET-1, pro-BNP, and various inflammatory markers will be checked before and 24 h after the procedure. It is our hypothesis that endothelial function will be better in the BNP treated patients compared to the NTG treated patients

ELIGIBILITY:
Inclusion Criteria:coronary artery disease -

Exclusion Criteria:CHF and/or reduced LV function, or renal failure with Creatinine >2mg%

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2005-07; Primary Completion 2012-04 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
FMD | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Mina Arinos, Principal Investigator — Ministry of Health, Israel
Locations (1):
- The Baruch Pade medical center, Poriya, Tiberias, Israel